CLINICAL TRIAL: NCT06768658
Title: A Randomized, Double-Blind, Placebo-Controlled Repeated Crossover Study to Evaluate the Safety and Tolerability of Intermittent Single Doses of TAK-951 in the Abortive Treatment of Subjects With Cyclic Vomiting Syndrome
Brief Title: A Study of TAK-951 in Participants With Cyclic Vomiting Syndrome (CVS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to business reasons prior to first subject dosed.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TAK-951-1501
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Nausea and Vomitting
Keywords: Drug Therapy
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (ABBA): Placebo + TAK-951 4 mg + TAK-951 4 mg + Placebo (Experimental): Participants will receive TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 1 (Period 1), followed by TAK-951 4 milligram (mg) (Treatment B), injection, subcutaneously, single dose, on Day 1 in CVS Episode 2 (Period 2), further followed by TAK-951 4 mg (Treatment B), injection, subcutaneously, single dose on Day 1 in CVS Episode 3 (Period 3), and further followed by TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 4 (Period 4). A washout period of at least 14 days will be maintained between each Period.
  Interventions: Drug: TAK-951; Drug: TAK-951 Placebo
- Sequence 2 (BAAB): TAK-951 4 mg + Placebo + Placebo + TAK-951 4 mg (Experimental): Participants will receive TAK-951 4 mg (Treatment B), injection, subcutaneously, single dose on Day 1 in CVS Episode 1 (Period 1), followed by TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 2 (Period 2), further followed by TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 3 (Period 3), and further followed by TAK-951 4 mg (Treatment B), injection, subcutaneously, single dose on Day 1 in CVS Episode 4 (Period 4). A washout period of at least 14 days will be maintained between each Period.
  Interventions: Drug: TAK-951; Drug: TAK-951 Placebo

INTERVENTIONS:
Drug: TAK-951 — TAK-951 subcutaneous injection.
Drug: TAK-951 Placebo — TAK-951 placebo-matching subcutaneous injection.

SUMMARY:
This is a study of TAK-951 in participants with cyclic vomiting syndrome (CVS).

The main aims of this study are as follows:

* To check for side effects from treatment with TAK-951.
* To learn how much TAK-951 participants can receive without getting side effects from it.
* To check how much TAK-951 stays in the blood over time to work out the best dose.
* The dose of TAK-951 will be checked to see how much stays in their blood over time.
* To see if it is possible to give treatment at home. Participants will be given TAK-951 injected just under the skin (subcutaneous or SC).

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements and is eligible for the study.
2. The participant or, when applicable, the participants' legally acceptable representative signs and dates a written or electronic, informed consent form and any required privacy authorization before the initiation of any study procedures.
3. The participant is male or female and aged 18 to 50 years, inclusive.
4. The participant has at least a 1-year history of CVS diagnosis based on the Rome IV diagnostic criteria.
5. The participant has had at least 4 CVS episodes over 6 months before screening during the last 12 months.
6. If taking eligible medications prescribed for the prophylaxis of CVS, the participant must be receiving a stable dose for at least 3 months before screening.
7. The participant is willing and able to exclusively use the protocol rescue medications if needed.
8. The participant has a stereotypic prodrome with onset less than or equal to (<=) 4 hours before CVS emetic events.
9. The participant has a body mass index (BMI) between 18 and 32 kilogram per square meter (kg/m^2), inclusive.
10. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use barrier method of contraception (example, condom with or without spermicide) from signing of informed consent throughout the duration of the study and for 30 days after last dose OR a surgically sterile female participant, or females of nonchildbearing potential with laboratory confirmation of postmenopausal status (that is, follicle-stimulating hormone levels greater than (>) 40 milli-international units per milliliter [mIU/mL]) or one of childbearing potential who is sexually active with a nonsterilized male partner agrees to use a highly effective method of contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose.

Exclusion Criteria:

1. The participant has participated in another interventional study within 4 weeks or 5 half-lives of the investigational study drug, whichever is longer, before the screening visit. The 4-week window will be derived from the date of the last study procedure and/or AE related to the study procedure in the previous study to the screening visit of the current study.
2. The participant has potentially received TAK-951 in a previous clinical study, or has previously completed, discontinued, or withdrawn from this study.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (example, spouse, parent, child, sibling) or is unable to provide consent (example, incapacity or potential duress or undue influence on informed consent process).
4. The participant has a history of significant multiple and/or severe allergies (example, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance (including medication-induced emesis) to prescription or nonprescription drugs or food, or allergic reactions to allowed rescue medication(s).
5. The participant has any condition or abnormality (including laboratory abnormalities), current or past, that, in the opinion of the investigator or medical monitor, would compromise the safety of the participant or interfere with or complicate the assessment of signs or symptoms of CVS.
6. The participant uses medical or recreational cannabis more than 3 days/week or its usage triggers nausea and/or vomiting.
7. The participant has a history of hypotension, autonomic instability, orthostatic hypotension (excluding in the context of concurrent dehydration), postural orthostatic tachycardia syndrome or a history or presence of 2 or more incidents of syncope within the last 5 years before screening.
8. Has a history of long corrected QT interval QTc, history of significant cardia arrhythmia, or a history or presence of:

   * A family history of unexplained sudden death or channelopathy; or
   * Brugada syndrome (that is, right bundle branch block pattern with ST-elevation in leads V1-V3); or
   * Second-degree atrioventricular block type 2, third degree atrioventricular block, prolonged QT interval with Fridericia correction method (QTcF) interval, hypokalemia, hypomagnesemia, or conduction abnormalities; or
   * Risk factors for Torsade de Pointes (example, heart failure, cardiomyopathy, or family history of Long QT Syndrome); or
   * Any clinically significant electrocardiogram (ECG) findings or medical history including: long or short QTcF (over 450 millisecond [msec] or less than 360 msec), bifascicular block or QRS greater than or equal to (>=120) msec or PR interval > 210 msec at screening; participants with QTcF >450 msec (up to 470 msec) taking chronic tricyclic antidepressants (>3 months) may be enrolled after consultation with the medical monitor; or o The participant has a documented history of sinus bradycardia (less than [<] 45 beats per minute [bpm]), sinoatrial block or sinus pause >=3 seconds, or sinus node dysfunction.
9. The participant has a history of other cardiovascular disease or cerebrovascular disease as assessed by the investigator including: essential hypertension requiring therapy or a history or presence of cerebrovascular disease such as cardiac valvulopathy, myocardial infarction, or stroke.
10. The participant has an average semirecumbent systolic blood pressure (SBP) < 95 or >140 or a diastolic blood pressure (DBP) <65 millimeter of mercury (mmHg) or >90 mm Hg at screening.
11. The participant has a screening average heart rate (HR) <55 or >100 bpm; athletic participants with a HR <55 bpm may be enrolled based upon the investigator's judgement provided that HR is >45 bpm and rhythm is sinus bradycardia.
12. The participant has orthostatic hypotension defined as a decrease in systolic blood pressure (BP) >=20 mmHg or a decrease in diastolic BP >=10 mmHg after approximately 3 minutes of standing when compared with BP from the semirecumbent position, at screening.
13. The participant has postural orthostatic tachycardia, defined as an increase of 30 bpm or HR >120 bpm after standing for approximately 3 minutes, at screening.
14. The participant is taking medications commonly associated with tachycardia, palpitations, hypotension, or QTc prolongation as potential adverse effects (example, beta blockers, nitrates, sildenafil).
15. The participant is taking medications prescribed for the prophylactic management of CVS with possible safety or tolerability interactions with TAK-951 as determined by the investigator(s). As above, chronic (>3 months) consistent dose of tricyclic antidepressants are allowed after consultation with the medical monitor if QTcF is <470. The use of prochlorperazine/or promethazine as a rescue medication is explicitly prohibited until >30 hours (5 half-lives of TAK-951) after investigational product administration.
16. The participant has a history of autonomic dysfunction.
17. The participant has active neoplastic disease or history of neoplastic disease within 5 years of screening visit (except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix that has been definitively treated with standard of care approaches) and has received treatment in the last 5 years.
18. The participant has a history of requiring emergency room/urgent medical treatment and intravenous fluid therapy for management of dehydration associated with clinically relevant hypotension for >2 CVS episodes in the last 6 months.
19. The participant has a history of other conditions associated with episodic emesis including: type 1 diabetes mellitus, type 2 diabetes mellitus, gastroparesis, gastrointestinal dysmotility, inflammatory bowel disease, eosinophilic esophagitis, rumination, severe functional dyspepsia, severe gastrointestinal reflux disease, large (>3 centimeter [cm]) hiatal hernia, or unrepaired intestinal malrotation.
20. The participant has taken opiate medications for more than 3 days in the last month.
21. The participant has a progressive neurological disorder or a structural disorder of the brain from birth, trauma or past infection.
22. The participant has an uncontrolled psychiatric disorder, to include history of suicide attempt, active major depressive disorder or severe panic disorder, or at the discretion of the investigator(s), for any clinically significant psychiatric history that would likely interfere with full participation in the study.
23. The participant has started a nonpharmacologic prophylactic approach (example, acupuncture, biofeedback, chiropractic methods) within 1 month before initiation of the treatment period.
24. The participant has a history of substance abuse.
25. The participant has a positive pregnancy test or plans to become pregnant during the study period.
26. The participant is a pregnant or lactating/nursing female.
27. The participant has a history of intolerance, hypersensitivity, or idiosyncratic reaction to TAK-951 (or any other glucose-dependent insulinotropic polypeptide [GIP] receptor agonist investigational products) or to any other ingredients of the investigational product.
28. The participant has a clinically unstable disease or condition.
29. The participant has any disease or condition that could compromise the function of those body systems as assessed by the investigator that could result in altered absorption, excess accumulation, or impaired metabolism or excretion of the test medications (example, mild, moderate or severe renal impairment [that is, creatinine clearance <90 milliliter per minute [mL/min] CrCL]) and/or altered hepatic function as assessed by the investigator (example, alanine aminotransferase [ALT] >2*the upper limit of normal [ULN], total bilirubin [TB]>1.5*ULN, alkaline phosphatase >1.5*ULN).
30. The participant has known or suspected active coronavirus disease 2019 infection as assessed by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- New Phase Research & Development, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/5d20c1506a0b46eb??page=1&idFilter=TAK-951-1501

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated by the sponsor due to business reasons, before any participant had been dosed in the study. One participant was screened but not dosed with study drug. No data were evaluated or collected for reporting in this study.
Groups:
- Sequence 1 (ABBA): Placebo + TAK-951 4 mg + TAK-951 4 mg + Placebo: Participants were to receive TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 1 (Period 1), followed by TAK-951 4 milligram (mg) (Treatment B), injection, subcutaneously, single dose, on Day 1 in CVS Episode 2 (Period 2), further followed by TAK-951 4 mg (Treatment B), injection, subcutaneously, single dose on Day 1 in CVS Episode 3 (Period 3), and further followed by TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 4 (Period 4). A washout period of at least 14 days was planned to be maintained between each Period.
- Sequence 2 (BAAB): TAK-951 4 mg + Placebo + Placebo + TAK-951 4 mg: Participants were to receive TAK-951 4 mg (Treatment B), injection, subcutaneously, single dose on Day 1 in CVS Episode 1 (Period 1), followed by TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 2 (Period 2), further followed by TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose on Day 1 in CVS Episode 3 (Period 3), and further followed by TAK-951 4 mg (Treatment B), injection, subcutaneously, single dose on Day 1 in CVS Episode 4 (Period 4). A washout period of at least 14 days was planned to be maintained between each Period.
Period: Overall Study
Arm/Group | Sequence 1 (ABBA): Placebo + TAK-951 4 mg + TAK-951 4 mg + Placebo | Sequence 2 (BAAB): TAK-951 4 mg + Placebo + Placebo + TAK-951 4 mg
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no data were evaluated and collected to be reported in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (ABBA): Placebo + TAK-951 4 mg + TAK-951 4 mg + Placebo | Sequence 2 (BAAB): TAK-951 4 mg + Placebo + Placebo + TAK-951 4 mg | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years] — Population: This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no data were evaluated and collected to be reported in this study.
Sex: Female, Male [unit: participants] — Population: This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no data were evaluated and collected to be reported in this study.
Ethnicity (NIH/OMB) [unit: participants] — Population: This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no data were evaluated and collected to be reported in this study.
Race (NIH/OMB) [unit: participants] — Population: This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no data were evaluated and collected to be reported in this study.
Region of Enrollment [unit: participants] — Population: This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no data were evaluated and collected to be reported in this study.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an adverse event (AE) with an onset that occurs after receiving study drug. An AE was defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study; it does not necessarily have to have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign (example, a clinically significant abnormal vital sign or laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it was considered related to the drug.
Time Frame: Up to end of study (up to 44 weeks)
Population: as for baseline characteristics
Groups:
- Placebo: Participants were to receive TAK-951 placebo-matching injection (Treatment A), subcutaneously, single dose, on Day 1 in CVS Episodes 1, 2, 3, or 4 (Periods 1, 2, 3 or 4). A washout period of at least 14 days was planned to be maintained between each Period.
- TAK-951 4 mg: Participants were to receive TAK-951 4 mg (Treatment B), injection, subcutaneously, single dose, on Day 1 in CVS Episodes 1, 2, 3, or 4 (Periods 1, 2, 3 or 4). A washout period of at least 14 days was planned to be maintained between each Period.
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Total Response
Description: Total response was defined as no emesis, no nausea (verbal rating scale [VRS] "none") and no need for rescue therapy before each time point. This was planned to be scored using a self-reported, 4-point VRS based on verbal responses of the participants to questions, where Score 0 - none; Score 1 - mild; Score 2 - moderate; and Score 3 - severe. Higher scores mean a worse outcome. Emesis was defined as vomiting (the forceful discharge of even the smallest amount of stomach contents) or retching (the same muscular movements as vomiting but without expulsion of stomach contents). Nausea was defined as the desire to vomit without the presence of expulsive muscular movements.
Time Frame: Within 2, 4, and 8 hours post-dose
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Absence of Emesis
Description: Absence of emesis was defined as no emesis and no need for rescue medication before each time point. Emesis was defined as vomiting (the forceful discharge of even the smallest amount of stomach contents) or retching (the same muscular movements as vomiting but without expulsion of stomach contents).
Time Frame: Within 2, 4, and 8 hours post-dose
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Absence of Significant Nausea
Description: Significant nausea was defined as a VRS greater than or equal to (>=) moderate. Absence of nausea was defined as VRS of "none" or "mild" and no need for rescue medication before the evaluation time point. This was planned to be scored using a self-reported, 4-point VRS based on verbal responses of the participants to questions, where Score 0 - none; Score 1 - mild; Score 2 - moderate; and Score 3 - severe. Higher scores mean a worse outcome. Nausea was defined as the desire to vomit without the presence of expulsive muscular movements.
Time Frame: Within 2, 4, and 8 hours post-dose
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Peak Nausea VRS Score in All Participants
Description: Nausea was defined as the desire to vomit without the presence of expulsive muscular movements. This was planned to be scored using a self-reported, 4-point VRS based on verbal responses of the participants to questions, where Score 0 - none; Score 1 - mild; Score 2 - moderate; and Score 3 - severe. Higher scores mean a worse outcome.
Time Frame: At 0, 1 and 2 hours post-dose
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Peak Nausea VRS Score in Participants Who Did Not Receive the Rescue Medication Before the Evaluation Timepoint
Description: as for outcome 5
Time Frame: At 4 and 8 hours post-dose
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Nausea VRS Score in All Participants
Description: as for outcome 5
Time Frame: At 1 and 2 hours post-dose
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Nausea VRS Score in Participants Who Did Not Receive the Rescue Medication Before the Evaluation Timepoint
Description: as for outcome 5
Time Frame: At 4 and 8 hours post-dose
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA)
Description: The ADA assessment was planned to be categorized as ADA negative, ADA positive and with low or high ADA titers. ADA negative was defined as participants who did not have a confirmed positive ADA status in any postbaseline assessment, and ADA positive as participants who had confirmed positive ADA status in any postbaseline assessment. High ADA titer was defined as participants who had at least 1 postbaseline ADA titer greater than (>) a cutoff planned to be determined based on the actual titer data, and Low ADA titer as participants whose postbaseline ADA titer numbers were all less than or equal to (<=) a cutoff planned to be determined based on the actual titer data.
Time Frame: Up to end of study (up to 44 weeks)
Population: as for baseline characteristics
Arm/Group | Placebo | TAK-951 4 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were not collected in this study.
Description: This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no death, serious adverse events (SAEs) and non-serious AE data were evaluated and collected to be reported in this study.
Arm/Group | Placebo | TAK-951 4 mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated early and only enrolled one participant that received no treatment. Due to concerns that the participant would be at risk of being re-identified and received no treatment, no data were evaluated and collected to be reported in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT06768658/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT06768658/SAP_001.pdf